CLINICAL TRIAL: NCT00986050
Title: A Comparison of Drug Eluting and Bare Metal Stents With or Without Abciximab in ST Segment Elevation Myocardial Infarction The Eindhoven Reperfusion Study
Brief Title: Comparison of Drug Eluting and Bare Metal Stents With or Without Abciximab in ST Elevation Myocardial Infarction
Acronym: DEBATER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Compusense Oegstgeest ( electronic randomization and CRF) (Unknown); CATHREINE ( data monitoring) (Unknown)
Responsible Party: Antoinette Spierings, CATHREINE
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CATHREINE-DEBATER 2006
Record Dates: First submitted 2009-09-09; First posted 2009-09-29 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2009-09

CONDITIONS: Acute Myocardial Infarction
Keywords: STEMI; DES; BMS; abciximab
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Abciximab; Drug-Eluting Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Bare metal stent (BMS) (Active Comparator)
  Interventions: Device: bare metal stent prokinetic, chrono, skylor or bluemedical
- Drug eluting stent (DES) (Active Comparator)
  Interventions: Device: drug eluting stent (sirolimus eluting) - CYPHER stent
- Abciximab (Active Comparator)
  Interventions: Drug: Abciximab
- No abciximab (No Intervention)

INTERVENTIONS:
Drug: Abciximab — Abciximab bolus 0,25mg/kg, 10-60 minutes before PCI. Infusion 0,125ug/kg/min for 12 hours after PCI.
  Other Names: reopro
  Arms: Abciximab
Device: bare metal stent prokinetic, chrono, skylor or bluemedical — bare metal stent in culprit artery in acute myocardial infarction
  Other Names: operator-dependent: prokinetic, chrono, skylor, bluemedical
  Arms: Bare metal stent (BMS)
Device: drug eluting stent (sirolimus eluting) - CYPHER stent — stent implantation in culprit artery in acute myocardial infarction
  Other Names: CYPHER stent
  Arms: Drug eluting stent (DES)

SUMMARY:
The DEBATER study is designed to determine the superiority of abciximab over no abciximab and to determine the superiority of drug eluting stents over bare metal stents in patients with acute myocardial infarction who undergo percutaneous coronary intervention.

DETAILED DESCRIPTION:
In patients with acute myocardial infarction primary PCI without prior thrombolytic therapy, is the treatment of choice.

The recommendation for routine stenting in PCI is based on 4 studies that have demonstrated the usefulness of bare metal stents in patients with STEMI. However this recommendation cannot be extrapolated (yet) to the use of drug eluting stents. Although DES have been used widely in unstable angina and in acute myocardial infarction, to date there are no evidence-based recommendations to support the routine use of DES in STEMI.

GPI have been studied extensively in patients with non-STsegment elevation myocardial infarctions (NSTEMI) with planned or performed PCI. In STEMI tirofiban and and eptifibatide are less well investigated, and only abciximab is recommended in primary PCI, but the long term benefits require more investigation. In PCI randomized controlled clinical trials (RCT's) abciximab consistently showed a significant reduction in the rate of myocardial infarction and the need for urgent revascularization. Abciximab has been evaluated in 5 RCT's in association with primary PCI. The pooled analysis for the clinical outcome at 30 days, demonstrate a significant reduction of death, re- infarction and target vessel revascularization (TVR), mainly due to a reduction of repeat intervention. The long-term benefits require more investigation.

The DEBATER trial is designed to answer the questions about the need for abciximab and about the use of DES in primary PCI.

ELIGIBILITY:
Inclusion Criteria:

* STEMI ≤ 12 hours (or STEMI equivalent).
* No contra - indications for primary PCI.
* No contra - indications for abciximab.
* Informed consent from the patient.

Exclusion Criteria:

* Contra - indication for primary PCI: History of peripheral/coronary artery disease that is inaccessible for angiography or PCI.
* Contra - indications for GPI: Ongoing bleeding, bleeding diathesis, cerebrovascular accident < 6 months, major surgery/trauma < 6 months, platelet count < 100.000 mm3 , intracranial arteriovenous malformation or neoplasm, malignant hypertension, INR >1.5, severe hepatic dysfunction
* Contra - indications for clopidogrel:

  * Severe liver dysfunction, pathological bleeding disorders such as peptic ulcer or intracranial bleeding.
  * Thrombolytic therapy < 24 hours.
  * Therapy with GPI < 24 hours.
  * Anticoagulation therapy.
* Co - morbid conditions with a predictable fatal outcome in the short run.
* No informed consent: refusal, coma, artificial respiration, impaired mentation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 907 (Actual)
Dates: Start 2006-01; Primary Completion 2008-05 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
target vessel failure | 30 days and one year

SECONDARY OUTCOMES:
Major adverse cardiac and cerebral adverse events ( MACCE) | 30 days and one year

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Michels, Principal Investigator — Catharina Ziekenhuis Eindhoven; Inge Wijnbergen, Principal Investigator — Catharina Ziekenhuis Eindhoven
Locations (1):
- Catharina ziekenhuis, Eindhoven, North Brabant, Netherlands

REFERENCES:
- [Background] Silber S, Albertsson P, Aviles FF, Camici PG, Colombo A, Hamm C, Jorgensen E, Marco J, Nordrehaug JE, Ruzyllo W, Urban P, Stone GW, Wijns W; Task Force for Percutaneous Coronary Interventions of the European Society of Cardiology. Guidelines for percutaneous coronary interventions. The Task Force for Percutaneous Coronary Interventions of the European Society of Cardiology. Eur Heart J. 2005 Apr;26(8):804-47. doi: 10.1093/eurheartj/ehi138. Epub 2005 Mar 15. PMID 15769784
- [Background] Montalescot G, Barragan P, Wittenberg O, Ecollan P, Elhadad S, Villain P, Boulenc JM, Morice MC, Maillard L, Pansieri M, Choussat R, Pinton P; ADMIRAL Investigators. Abciximab before Direct Angioplasty and Stenting in Myocardial Infarction Regarding Acute and Long-Term Follow-up. Platelet glycoprotein IIb/IIIa inhibition with coronary stenting for acute myocardial infarction. N Engl J Med. 2001 Jun 21;344(25):1895-903. doi: 10.1056/NEJM200106213442503. PMID 11419426
- [Background] Schomig A, Schmitt C, Dibra A, Mehilli J, Volmer C, Schuhlen H, Dirschinger J, Dotzer F, ten Berg JM, Neumann FJ, Berger PB, Kastrati A; Intracoronary Stenting and Antithrombotic Regimen-Rapid Early Action for Coronary Treatment Study Investigators. One year outcomes with abciximab vs. placebo during percutaneous coronary intervention after pre-treatment with clopidogrel. Eur Heart J. 2005 Jul;26(14):1379-84. doi: 10.1093/eurheartj/ehi174. Epub 2005 Feb 25. PMID 15734767
- [Derived] Wijnbergen I, Helmes H, Tijssen J, Brueren G, Peels K, van Dantzig JM, Van' t Veer M, Koolen JJ, Pijls NH, Michels R. Comparison of drug-eluting and bare-metal stents for primary percutaneous coronary intervention with or without abciximab in ST-segment elevation myocardial infarction: DEBATER: the Eindhoven reperfusion study. JACC Cardiovasc Interv. 2012 Mar;5(3):313-22. doi: 10.1016/j.jcin.2011.11.009. PMID 22440498